CLINICAL TRIAL: NCT07353307
Title: To Evaluate the Efficacy, Safety and Pharmacokinetics of TRD303 Solution for Postoperative Analgesia After Abdominal Surgery in a Multicenter, Randomized, Double-blind, Placebo-positive Controlled Phase Ⅲ Clinical Trial
Brief Title: A Clinical Trial Evaluating the Efficacy, Safety, and Pharmacokinetic Profile of TRD303 for Postoperative Analgesia After Abdominal Surgery in China.
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Yingyong Zhou,MD,PhD, PhD, The Third Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRD303-Ⅲ -02
Record Dates: First submitted 2025-12-29; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Pain After Abdominal Surgery
MeSH Terms: interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TRD303 group (Experimental): Before the surgical incision was closed, TRD303 solution was applied to the incision wound.
  Interventions: Drug: TRD303 solution
- Positive control group (Active Comparator): Before the surgical incision was closed, 0.5% ropivacaine hydrochloride was injected into the incision wound
  Interventions: Drug: Ropivacaine hydrochloride
- Placebo control group (Placebo Comparator): Before the surgical incision was closed, the incision wound was infiltrated with 0.9% sodium chloride injection
  Interventions: Drug: 0.9 % sodium chloride

INTERVENTIONS:
Drug: TRD303 solution — After the peritoneum was sutured, the final irrigation and suction were performed, and the wound was smeered with TRD303 solution after incision injection before the surgical incision was sutured. The injection volume of the main incision was 2.5mL (±0.5mL was allowed according to the actual situation of the incision). For surgery involving multiple incisions, the secondary incisions were administered according to the number of incisions per unit, and the drug administration volume of each incision was 0-0.5 mL (0mL≤ administration volume ≤0.5mL).
  Other Names: Before the surgical incision was closed, TRD303 solution was applied to the incision wound.
  Arms: TRD303 group
Drug: Ropivacaine hydrochloride — After the completion of peritoneal suture, final irrigation and aspiration, 0.5% ropivacaine hydrochloride was injected locally around the incision before the surgical incision was closed. If there was residual drug solution after the administration of the primary incision, the residual drug solution was used to the secondary incision infiltration, and a total of 30mL was given.
  Arms: Positive control group
Drug: 0.9 % sodium chloride — After the suture of the peritoneum, final irrigation and aspiration, 0.9% sodium chloride injection was injected locally around the incision before the suture of the surgical incision. If there was residual drug solution after the administration of the primary incision, the residual drug solution was used to the secondary incision infiltration, and a total of 30mL was given.
  Arms: Placebo control group

SUMMARY:
A multicenter, randomized, double-blind, placebo-positive, parallel-controlled, phase Ⅲ clinical trial of the efficacy, safety and pharmacokinetics of TRD303 solution for postoperative analgesia in patients undergoing abdominal surgery was conducted. The primary objective was to evaluate the efficacy of TRD303 solution for postoperative analgesia after abdominal surgery. The secondary objective was to evaluate the safety and pharmacokinetic profile of TRD303 solution for postoperative analgesia after abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the purpose and significance of this study, voluntarily participate in this study, voluntarily sign the informed consent, and voluntarily abide by the process of this study;
2. 18 years old ≤ age ≤80 years old, regardless of gender; 18.0kg/m2≤BMI≤30.0kg/m2, ≥50.0kg for men and ≥45.0kg for women;

4. American Society of Anesthesiologists (ASA) grade I-II (Appendix 1); (5) Elective abdominal surgery under general anesthesia, including laparoscopic or open surgery, and the length of the main incision is expected to be between 7±2cm (including the boundary value at both ends); 6. Can understand the research process and the use of various scales involved in this study, and can effectively communicate with researchers.

Exclusion Criteria:

1. Those who are known to have allergies or contraindications to ropivacaine or other amide local anesthetics, inactive ingredients of the investigational drug, or other drugs that may be used during the trial, and who are judged by the investigator to be unsuitable for the trial;
2. Use of the following drugs for less than 5 half-lives before randomization (according to the actual drug instructions, the half-life is unknown, or eluted according to 48 hours), including but not limited to: Class III antiarrhythmic drugs, glucocorticoids (systemic), anticonvulsants, sedative-hypnotic drugs, anxiolytic drugs, antidepressant drugs, CYP1A2 enzyme inhibitor, sedative drugs (except those used according to the protocol), analgesic drugs (except those used according to the protocol), the specific types refer to the list of prohibited drugs; Use of Chinese herbal medicine with definite analgesic effect assessed by investigators within 7 days before randomization;
3. Participants who planned to use hyperthermic perfusion, intraperitoneal chemotherapy, physical therapy, or other concomitant therapies during the treatment period that the investigator judged might affect postoperative pain;
4. patients who underwent abdominal surgery within 1 year before signing ICF;
5. patients who planned to undergo surgery at other sites during the study period;
6. Combined with other pain conditions that may confound the evaluation of postoperative pain according to the investigator;
7. Participants with a history of congenital or idiopathic methemoglobinemia or glucose-6-phosphate dehydrogenase deficiency;
8. Previous and/or family history of malignant hyperthermia;
9. Participants with poorly controlled blood pressure during screening (systolic blood pressure ≥160mmHg or ≤90 mmHg while sitting during screening, and/or diastolic blood pressure ≥100 mmHg or ≤60mmHg during screening, excluding abnormal blood pressure during anesthesia), whose abnormalities were judged by the investigator to be clinically significant and increase perioperative risk;
10. Heart rate < 50 beats/min or heart rate > 100 beats/min during screening (excluding abnormal heart rate during anesthesia), and the abnormal heart rate was judged by the investigator to be clinically significant; QTcF > 450ms in men and > 470ms in women [QTcF=QT/ (RR^0.33)]; Or a history of severe arrhythmias such as atrioventricular block of degree II or higher, or cardiac insufficiency;
11. Patients with severe liver, kidney, cardiovascular, cerebrovascular, or metabolic diseases judged by the investigator to be unsuitable for the trial;
12. Patients with advanced malignant tumors who were judged by the investigators to be not suitable for participating in the trial;
13. Patients with a history of mental diseases (such as schizophrenia, depression, etc.), dementia, migraine, or epilepsy, who were judged by the investigator to be unfit for the trial;
14. Patients with skin infection, ulceration or scar constitution around the incision, judged by the investigator to be not suitable for the trial;
15. Participants with a history of psychoactive and narcotic drug abuse, drug use, and heavy drinking (i.e., drinking an average of more than 2 units of alcohol per day (1 unit =360mL of beer or 45mL of 40% liquor or 150 ml of wine) in the year before randomization;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Area under curve (AUC) of the pain intensity-time during 0-72h at rest | From administration until 72 hours after administration
  Area under the resting pain intensity time curve (AUC0-72h) during 0-72 hours after administration

SECONDARY OUTCOMES:
Area under the pain intensity time curve at rest | From administration until 4 hours, 6 hours, 12 hours, 24 hours, 48 hours after administration, from 24 hours to 48 hours after administration, from 48 hours to 72 hours after administration
  The area under the pain intensity time curve (AUC0-4h, AUC0-6h, AUC0-12h, 0-24h, AUC0-48h, AUC24-48h, AUC48-72h) in resting state during 0-4h, 0-6h, 0-12h, 0-24h, 0-48h, 24-48h, and 48-72h after the completion of administration.
Area under the pain intensity time curve during exercise | From the time of administration to 12 hours, 24 hours, 48 hours, 72 hours after administration, from 24 hours to 48 hours after administration, from 48 hours to 72 hours after administration
  Area under the pain intensity time curve (AUC0-12h, AUC0-24h, AUC0-48h, AUC0-72h, AUC24-48h, AUC48-72h) during exercise during 0-12h, 0-24h, 0-48h, 0-72h, 24-48h, and 48-72h after the completion of administration.
Time of first morphine rescue analgesia | From administration until 72 hours after administration
  The time from the completion of administration to the first morphine rescue analgesic treatment
Cumulative use of rescue analgesics during each period | From the time of administration to 4 hours, 6 hours, 12 hours, 24 hours, 48 hours, 72 hours after administration
  Cumulative amount of rescue analgesics used during 0-4h, 0-6h, 0-12h, 0-24h, 0-48h, and 0-72h after completion of administration
The number of rescue analgesia in each period | From the time of administration to 4 hours, 6 hours, 12 hours, 24 hours, 48 hours, 72 hours after administration
  The cumulative number of rescue analgesics used during 0-4h, 0-6h, 0-12h, 0-24h, 0-48h, and 0-72h after the completion of administration
Proportion of rescue analgesia in each period | From the time of administration to 4 hours, 6 hours, 12 hours, 24 hours, 48 hours, 72 hours after administration
  Proportion of participants who used rescue analgesics within 0-4h, 0-6h, 0-12h, 0-24h, 0-48h, and 0-72h after administration

OTHER OUTCOMES:
Maximum Plasma Concentration (Cmax) of TRD303 | From administration until 72 hours after administration
  Maximum plasma concentration of TRD303 after Administration
Area under curve (AUC) of the plasma concentration-time during 0-t (t=0 to 48h) | From administration until time t (t=0 to 48h) after administration
  The area under the drug concentration-time curve from the start of drug administration to time t (AUC0-t, t=0 to 48h)
Area under curve (AUC) of the plasma concentration-time during 0-∞ (AUC0-∞) | From administration until 7 days post-administration, continuing until all prototype drugs were completely eliminated.
  Total area under the curve from administration until all the prototypic drugs were eliminated (AUC0-∞)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Sichuan Provincial People's Hospital, Sichuan

IPD SHARING:
Plan to Share IPD: No